CLINICAL TRIAL: NCT04633681
Title: Acute and Repeated Impact of Sweeteners and Sweetness Enhancers on Food Behaviour, Physiology & Health (SWEET Work Package 2 Phase 2)
Brief Title: Impact of Sweeteners on Behaviour, Physiology & Health
Acronym: SWEET-WP2-P2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: University of Navarra (Other); University of Liverpool (Other); Københavns Universitet (Other); Centre de Recherche en Nutrition Humaine Rhone-Alpe (Other); University of Surrey (Other); Bioatriki Healthcare Group (Unknown)
Responsible Party: Principal Investigator, Dr Graham Finlayson, Professor, University of Leeds
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 774293-WP2-P2
Record Dates: First submitted 2020-10-30; First posted 2020-11-18 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Eating Behavior
Keywords: appetite; food preferences; sweeteners; sweetness enhancers
MeSH Terms: conditions — Feeding Behavior; Food Preferences | interventions — Sweetening Agents

STUDY DESIGN:
Intervention Model Description: Double-blind, within-subjects, cross-over trial
Who Masked: Participant, Investigator
Masking Description: Double blind study. Neither the participant nor the investigator will be aware of the coding of food products used in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Cake matrix (Experimental): 3 phases of 2-week daily consumption of cake product containing 1) sucrose, 2) Neotame 1, 3) Stevia Reb M. Randomised cross-over with 2-week wash-out between phases.
  Interventions: Dietary Supplement: Sweetener and sweetness enhancer consumption
- Biscuit matrix (Experimental): 3 phases of 2-week daily consumption of biscuit product containing 1) sucrose, 2) Neotame 1, 3) Stevia Reb M. Randomised cross-over with 2-week wash-out between phases.
  Interventions: Dietary Supplement: Sweetener and sweetness enhancer consumption
- Yoghurt matrix (Experimental): 3 phases of 2-week daily consumption of yoghurt product containing 1) sucrose, 2) sweetener blend 1, 3) sweetener blend 2. Randomised cross-over with 2-week wash-out between phases.
  Interventions: Dietary Supplement: Sweetener and sweetness enhancer consumption
- Chocolate matrix (Experimental): 3 phases of 2-week daily consumption of chocolate product containing 1) sucrose, 2) sweetener blend 1, 3) sweetener blend 2. Randomised cross-over with 2-week wash-out between phases.
  Interventions: Dietary Supplement: Sweetener and sweetness enhancer consumption
- Cereal matrix (Experimental): 3 phases of 2-week daily consumption of cereal product containing 1) sucrose, 2) sweetener blend 1, 3) sweetener blend 2. Randomised cross-over with 2-week wash-out between phases.
  Interventions: Dietary Supplement: Sweetener and sweetness enhancer consumption
- Universal Eating Monitor study (Experimental): A sub-group of the yoghurt matrix will be selected for assessment of eating rate and microstructure of feeding using Universal Eating Monitors.
  Interventions: Dietary Supplement: Sweetener and sweetness enhancer consumption
- fMRI study (Experimental): A sub-group of the chocolate matrix will be selected for assessment of neural activation to images of food using fMRI.
  Interventions: Dietary Supplement: Sweetener and sweetness enhancer consumption

INTERVENTIONS:
Dietary Supplement: Sweetener and sweetness enhancer consumption — Two-week consumption of combinations of different sweetener and sweetness enhancer blends in reformulated food products compared to sucrose containing product.

SUMMARY:
This study aims to evaluate the acute (1-day) and repeated (2-week) effects of combinations of Sweeteners & Sweetness Enhancer blends on metabolic, sensory, neuro-behavioural and microbiota-mediated processes involved in satiety, consumer preferences and health.

DETAILED DESCRIPTION:
This protocol has the overall objective to evaluate the acute (short-term, 1 day) and repeated (medium-term, 2 week) effects of combinations of sweeteners and sweetness enhancers (S&SEs) on metabolic, sensory, neuro-behavioural and microbiota-mediated processes involved in satiety, consumer preference and health, and to explore mechanistic processes, genetic background, safety issues and consumer perspectives.

There are 5 products being tested in 3 different formulations (sucrose-sweetened control vs 2 reformulated with S&SE). Each product will be tested at 2 intervention sites in double-blind cross-over trials with 48 subjects (24 per site) tested per product. Therefore a total of 240 subjects will take part across the 5 intervention sites (Navarra, Leeds, Liverpool, Copenhagen, Lyon).

Using identical procedures each trial will consist of 2 Clinical Investigation Days (CIDs) scheduled 12 days apart for each of the 3 product formulations. A 2-week wash-out period will be given between formulations.

The total duration of WP2 Phase 2 is 12 months, including a 5-month duration for each cross-over trial.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 25 to 35 kg/m2
* Use of contraceptive methods or not planning to become pregnant for the duration of the study (women only)
* Regular consumption of sugar-containing foods and willing to consume sugar and artificially-sweetened food products.
* Liking of the intervention foods defined by a response of Yes for the product during the pre-screening interview and a score of 40% or above on the Liking Visual Analogue Scale for the sucrose-sweetened control product.
* Able to participate on the Clinical Investigation Days during normal working hours.
* Healthy as determined from the self-reported medical history or when a clinical condition exists, when this is considered to be irrelevant (i.e. not influencing study outcomes) for the study by the study medical doctor.
* Consuming breakfast regularly (at least 5 days per week).
* Able to understand and be willing to sign the informed consent form, and to follow all the study procedures and requirements.
* Capacity to store at-home intervention quantity of intervention product

Exclusion Criteria:

* Blood donation < 3 month prior to study or for full duration of the study.
* Food allergy, intolerance, restriction or avoidance of any of the study foods (e.g. veganism) or history of anaphylactic reaction to any food.
* Likelihood for disordered eating defined as a score ≥20 on the Eating Attitudes Test.
* Currently dieting to lose weight.
* Having lost or gained >4.5 kg in the last 3 months.
* Smoking or having quit <3 months prior to study.
* Habitually consuming >14 units/week of alcohol in women or >21 units/week in men in the last 3 months.
* Performing >10 h of intense physical activity per week in the last 3 months.
* Night or late shift work (ending later than 11 pm on a permanent basis). Rotational shift work allowed if can attend on days that do not follow a late/night shift.
* Self-reported use of drugs of abuse within the previous 12 months.
* Pregnancy, lactation (women only)
* Persons who do not have access to either (mobile) phone or internet (this is necessary when being contacted by the study personnel during the study).
* Insufficient communication in the national language.
* Proven or suspected inability, physically or mentally, to comply with the procedures required by the study protocol as evaluated by the daily study manager, site-PI, PI or clinical responsible. This includes volunteers for which insufficient collaboration may be foreseen.
* Subject's general condition contraindicates continuing in the study as evaluated by the daily study manager, site-PI, PI or responsible clinician.
* Simultaneous participation in other relevant clinical intervention studies.
* Previous university or college training related to eating behaviour research.
* Self-reported eating disorders.
* Diagnosed anaemia.
* Diagnosed diabetes mellitus.
* Abnormal G.I. function or structure such as malformation, angiodysplasia, active peptic ulcer.
* Active inflammatory bowel disease, celiac disease, chronic pancreatitis or other disorder potentially causing malabsorption.
* History of G.I. surgery with permanent effect (i.e. surgical treatment of obesity).
* Medical history of Cardiovascular Disease (e.g. current angina; myocardial infarction or stroke within the past 6 months; heart failure; symptomatic peripheral vascular disease).
* Significant liver disease, e.g. cirrhosis (fatty liver disease allowed).
* Malignancy which is currently active or in remission for less than five years after last treatment (local basal and squamous cell skin cancer allowed).
* Thyroid diseases, except those on Levothyroxine treatment of hypothyroidism if the person has been on a stable dose for at least 3 months.
* Psychiatric illness (e.g. major depression, bipolar disorders).
* Use currently or within the previous 3 months of prescription or over the counter medication that has the potential of affecting appetite, satiety or body weight incl. food supplements. Except: low dose antidepressants if they, in the judgement of the daily study manager, site-PI, PI or clinical responsible, do not affect weight or following the study protocol. Levothyroxine for treatment of hypothyroidism is allowed if the person has been on a stable dose for at least 3 months.
* Cholesterol lowering medication, if the dose has changed during the last 3 months (i.e. the medication is allowed if the participant has been on a stable dose for at least 3 months).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 175 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Composite Appetite Sensations Incremental Area Under the Curve | Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Incremental area under the curve (iAUC) for composite appetite sensations in response to each product.
  During each of the Clinical Investigation Days iAUC composite appetite will be measured 180 minutes post intake.
  The following sensations of appetite will be used in the composite measure:
  * hunger
  * fullness
  * desire to eat
  * prospective consumption
  Minimum value 0 Maximum value 100 Higher scores mean worse outcome

SECONDARY OUTCOMES:
Leeds Food Preference Questionnaire (LFPQ) Explicit Liking | Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Change in explicit liking for foods at 15 min post intake Minimum value -100 Maximum value 100 Higher scores mean worse outcome
Leeds Food Preference Questionnaire (LFPQ) Implicit Wanting | Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Change in implicit wanting for foods at 15 min post intake Minimum value -100 Maximum value 100 Higher scores mean worse outcome
Leeds Food Preference Questionnaire (LFPQ) Relative preference | Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Change in relative preference for foods at 15 min post intake Minimum value -48 Maximum value 48 Higher scores mean worse outcome
Leeds Food Preference Questionnaire (LFPQ) Explicit wanting | Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Change in explicit wanting for foods at 15 min post intake Minimum value -100 Maximum value 100 Higher scores mean worse outcome
Control of Eating Questionnaire (CoEQ): Craving Control | Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Craving Control examined in a fasted state. Minimum value 0 Maximum value 100 Higher scores mean better outcome
Control of Eating Questionnaire (CoEQ): Craving for Sweet | Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Craving for Sweet examined in a fasted state. Minimum value 0 Maximum value 100 Higher scores mean worse outcome
Control of Eating Questionnaire (CoEQ): Craving for Savoury | Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Craving for Savoury examined in a fasted state. Minimum value 0 Maximum value 100 Higher scores mean worse outcome
Control of Eating Questionnaire (CoEQ): Positive Mood | Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Positive Mood examined in a fasted state. Minimum value 0 Maximum value 100 Higher scores mean better outcome
Blood Glucose Incremental Area Under the Curve | Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Incremental area under the curve for blood glucose concentrations in response to each product (120 min post intake).
Blood Insulin Incremental Area Under the Curve | Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Incremental area under the curve for blood insulin concentrations in response to each product (120 min post intake).
Cephalic and intestinal satiety biomarkers: Glucagon-like peptide-1 (GLP-1) | Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Incremental area under the curve for blood GLP-1 concentrations in response to each product (120 min post intake).
Cephalic and intestinal satiety biomarkers: Ghrelin | Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Incremental area under the curve for blood Ghrelin concentrations in response to each product (120 min post intake).

OTHER OUTCOMES:
Body composition: fat mass (kg) | Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Anthropometry marker fat mass
Body composition: fat-free mass (kg) | Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Anthropometry marker fat-free mass
Body weight (kg) | Fasting during each Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Anthropometry marker body weight
Standing height (cm) | Measured in a fasting state during screening day only
  Anthropometry marker standing height
Waist circumference (cm) | Fasting during each Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Anthropometry marker waist circumference
Body composition, body weight, height, waist and hip circumference | Fasting during each Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Anthropometry marker hip circumference
Sweet taste receptor polymorphism prevalence | Clinical Investigation Day 1 only in a fasted state
  Blood DNA analysis for sweet taste receptor polymorphism prevalence
Consumers' Perspectives Questionnaire on sweeteners | Fasted state on screening day only (Day 0)
  Psychological health drivers (perceptions) of sweetener consumption
Gut microbiota profile (diversity and ratio) | Collected the day before each Clinical Investigation Day for the yoghurt food matrix.
  Gut microbiota measured from fecal samples during clinical investigation days in yoghurt matrix only
Brain activity (fMRI) | Clinical Investigation Day 1 and Clinical Investigation Day 6 immediately before and immediately after consumption of the chocolate food matrix.
  Neural activation to chocolate matrix only
Meal eating behaviour and microstructure: Eating rate | Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Eating rate using the Universal Eating Monitor in yoghurt matrix only
Meal eating behaviour and microstructure: Bite count | Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Bite count using the Universal Eating Monitor in yoghurt matrix only
Urinary S&SEs biomarkers | Collected the day before each Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Biomarkers of S&SE quality measured from urine samples
Eating behaviour traits: Three factor eating questionnaire Restraint subscale | Fasted state on screening day only (Day 0)
  Restraint eating behaviour trait measured by the Three Factor Eating Questionnaire.
  Minimum value 0 Maximum value 21 Higher scores mean worse outcome
Eating behaviour traits: Three factor eating questionnaire Hunger subscale | Fasted state on screening day only (Day 0)
  Hunger eating behaviour trait measured by the Three Factor Eating Questionnaire.
  Minimum value 0 Maximum value 14 Higher scores mean worse outcome
Eating behaviour traits: Three factor eating questionnaire Disinhibition subscale | Fasted state on screening day only (Day 0)
  Disinhibition eating behaviour trait measured by the Three Factor Eating Questionnaire.
  Minimum value 0 Maximum value 16 Higher scores mean worse outcome
Eating behaviour traits: Binge Eating Scale | Fasted state on screening day only (Day 0)
  Binge Eating measured by the Binge Eating Scale
  Minimum value 0 Maximum value 46 Higher scores mean worse outcome
Habitual intake of sweet foods | Fasted state on screening day only (Day 0)
  Short sugar Food Frequency Questionnaire (short sFFQ)
Perception and evaluation of the clinical trial | Clinical Investigation Day 6
  End of study survey
24-h Dietary recall: Self-reported energy intake | Next day after each Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Interview to know what the volunteers ate during the 24h following each probe day
24-h Dietary recall: Energy compensation after intake of intervention products | Next day after each Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Interview to know what the volunteers ate during the 24h following each probe day accounting for the energy contained in the intervention food products
Expected satiety | Immediately before consuming food product during each Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Single-item Visual Analogue Scale assessing expected satiety from the intervention food products Minimum value 0 Maximum value 100 Higher scores mean better outcome
Sensory-specific satiety | Immediately before and immediately after consuming food product during each Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Single-item Visual Analogue Scale assessing sensory-specific satiety from the intervention food products Minimum value 0 Maximum value 100 Higher scores mean better outcome
Thirst Incremental Area Under the Curve | Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Incremental area under the curve (iAUC) for thirst in response to each product.
  During each of the Clinical Investigation Days iAUC thirst will be measured 180 minutes post intake using visual analogue scale.
  Minimum value 0 Maximum value 100 Higher scores mean worse outcome
Nausea Incremental Area Under the Curve | Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Incremental area under the curve (iAUC) for nausea in response to each product.
  During each of the Clinical Investigation Days iAUC nausea will be measured 180 minutes post intake using visual analogue scale.
  Minimum value 0 Maximum value 100 Higher scores mean a worse outcome.
Bloating Incremental Area Under the Curve | Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Incremental area under the curve (iAUC) for bloating in response to each product.
  During each of the Clinical Investigation Days iAUC bloating will be measured 180 minutes post intake using visual analogue scale.
  Minimum value 0 Maximum value 100 Higher scores mean worse outcome
Cephalic and intestinal satiety biomarkers: Pancreatic polypeptide (PP) | During each of the probe day visits blood pancreatic polypeptide (PP) will be measured at baseline, and 5, 10, 30 minutes after consuming the product. Each visit will be separated by 12 days of daily consumption of the product.
  Incremental area under the curve for blood PP concentrations in response to each product (120 min post intake).
Lipaemia: triglycerides | Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Incremental area under the curve for blood triglyceride concentrations in response to each product (120 min post intake).
Lipaemia: Cholesterol (total) | Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Incremental area under the curve for blood cholesterol (total) concentrations in response to each product (120 min post intake).
Lipaemia: Cholesterol (HDL) | Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Incremental area under the curve for blood cholesterol (HDL) concentrations in response to each product (120 min post intake).
Lipaemia: Cholesterol (LDL) | Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Incremental area under the curve for blood cholesterol (LDL) concentrations in response to each product (120 min post intake).
Liver function: Alanine aminotransferase (ALT) | Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Mean of liver function marker (ALT) concentrations in response to each product (120 min post intake).
Liver function: Aspartate aminotransferase (AST) | Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Mean of liver function marker (AST) concentrations in response to each product 120 min post intake.
Liver function: Gamma-Glutamyl Transpeptidase (GGT) | Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Mean of liver function marker (GGT) concentrations in response to each product 120 min post intake.
Liver function: Fatty Liver index | Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Mean of liver function marker (FL index) concentrations in response to each product 120 min post intake.
Liver function: Triglyceride index | Clinical Investigation Day 1, 2, 3, 4, 5, 6
  Mean of liver function marker (TyG index) concentrations in response to each product 120 min post intake.
HbA1c | Measured in a fasting state during Clinical Investigation Day 1 and 6 only
  Fasting HbA1c blood concentrations
24 hour Gastrointestinal side effects | Up to 24 hours after each Clinical Investigation Day and from Clinical Investigation Day 1, 2, 3, 4, 5, 6 during the 3 at home intervention periods up to 12 days
  GI side effects reported in a booklet to know if the volunteers experience side effects during the intervention periods
Adverse events | Up to 24 hours after each Clinical Investigation Day and from Clinical Investigation Day 1, 2, 3, 4, 5, 6 during the 3 at home intervention periods up to 12 days
  Adverse event reported in a booklet to know if the volunteers experience side effects during the intervention periods

CONTACTS AND LOCATIONS:
Locations (5):
- University of Copenhagen, Copenhagen, Denmark
- CRNH-RA, Lyon, France
- University of Navarra, Pamplona, Spain
- United Kingdom (2):
  - University of Leeds, Leeds, West Yorkshire
  - University of Liverpool, Liverpool

REFERENCES:
- [Derived] Gibbons C, O'Hara B, O'Connor D, Hardman C, Wilton M, Harrold JA, Almiron-Roig E, Navas-Carretero S, Hodgkins CE, Nazare JA, Alligier M, Martinez JA, Scott C, Kjolbaek L, Normand M, Rannou C, Blaak EE, Feskens E, Moshoyiannis H, Raben A, Halford JCG, Beaulieu K, Finlayson G. Acute and repeated impact of sweeteners and sweetness enhancers in solid and semi-solid foods on appetite: protocol for a multicentre, cross-over, RCT in people with overweight/obesity - the SWEET Project. BMJ Open. 2022 Dec 23;12(12):e063903. doi: 10.1136/bmjopen-2022-063903. PMID 36564114